CLINICAL TRIAL: NCT01001897
Title: A Randomized Control Trial of Misoprostol vs. Placebo for Cervical Preparation in IUD Insertion for Nulliparous Women
Brief Title: Use of Misoprostol for Intrauterine Device (IUD) Insertion in Nulliparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Pam Lotke, Principal Investigator, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 09004201
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Contraception
Keywords: IUD insertion; nulliparous women; contraception
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- misoprostol (Experimental): 400 micrograms of misoprostol inserted buccally or vaginally prior to IUD insertion
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): Troches identical to experimental drug inserted buccally or vaginally prior to IUD insertion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — 400 micrograms of misoprostol or placebo inserted buccally or vaginally prior to IUD insertion
  Arms: misoprostol
Drug: Placebo — 400 micrograms of misoprostol or placebo inserted buccally or vaginally prior to IUD insertion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if the use of misoprostol can make it easier for a provider, and less painful for a woman, to place an IUD if she has never had a child before.

DETAILED DESCRIPTION:
IUD's are a tremendously effective long acting, reversible method of contraception, and they require little participation from the woman after insertion. Despite these benefits, few women in the US use an IUD. Education is important so that both providers and women understand that IUD's are safe and effective in women even if they have never had a child. Insertion of an IUD in nulliparous patients can be more difficult and uncomfortable. The purpose of this study is to see if use of misoprostol prior to IUD placement in nulliparous women can make it easier and less painful. The goal is that more information on the feasibility and ease of IUD insertion will make it more accessible to more women. The findings from this trial will be used in a prospective meta analysis on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous, no prior pregnancy beyond 14 week
* Over 18 years of age
* Negative pregnancy test

Exclusion Criteria:

* current pregnancy or pregnancy within 6 weeks
* current cervicitis or PID (active or within 3 months)
* undiagnosed abnormal uterine bleeding
* allergy to copper/ Wilson's disease (for Paragard)
* cervical or uterine cancer
* uterine anomaly altering uterine cavity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is worst perceived pain during the IUD insertion procedure, on a 100 mm visual analogue scale | after IUD insertion

SECONDARY OUTCOMES:
Need to use adjuvant measures for IUD placement, such as dilation, ultrasound guidance, anesthesia | during IUD insertion
Side effects of medications | prior to IUD insertion
Provider perceived ease of insertion on a 100 mm visual analogue scale | after IUD insertion
Acceptability of wait time prior to IUD placement | 1 week after IUD insertion
Procedure complications | Up to 1 month after IUD placement
Acceptability of total IUD placement process, would you recommend this to a friend? | 1 week and 1 month after IUD insertion

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UPH-Kino multispecialty clinic, Tucson, Arizona
  - University Medical Center Ob/Gyn clinic 8OPC, Tucson, Arizona

REFERENCES:
- [Derived] Espey E, Singh RH, Leeman L, Ogburn T, Fowler K, Greene H. Misoprostol for intrauterine device insertion in nulliparous women: a randomized controlled trial. Am J Obstet Gynecol. 2014 Mar;210(3):208.e1-5. doi: 10.1016/j.ajog.2013.11.018. Epub 2013 Nov 8. PMID 24215850
- [Derived] Turok DK, Espey E, Edelman AB, Lotke PS, Lathrop EH, Teal SB, Jacobson JC, Simonsen SE, Schulz KF. The methodology for developing a prospective meta-analysis in the family planning community. Trials. 2011 Apr 29;12:104. doi: 10.1186/1745-6215-12-104. PMID 21527040